CLINICAL TRIAL: NCT05485389
Title: The Effect of Simulation Based Learning on Improve Positive Attitudes and Individualized Care Perceptions of Nurses Towards Elderly Patient
Brief Title: The Effect of Simulation to Improve of Nurse's Attitudes Towards Elderly Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1122334455
Record Dates: First submitted 2022-07-30; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Simulation Training; Elderly; Nursing Care
Keywords: Simulation based learning; Elderly patient; nursing attitudes; Individualized care

STUDY DESIGN:
Intervention Model Description: pre-test and post-test semi-experimental design
Masking Description: The nurses included in the study were named as participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): At the beginning, knowledge test, individualized care perception and attitude scale to the elderly will be applied to the participants in the pre-test. Then, 6-hour theoretical course on the care of the elderly patient will be given to the participants included in the study. After the theoretical course, the knowledge test will be re-applied. After that, experience will be provided within the scope of first, second and third level simulation-based learning, one week apart. After the simulation experiences knowledge test, individualized care perception and attitude scale to the elderly will be applied to the participants in the post-test 1. Post-tests will be administered in the first (Post-test 2) and third (Post-test 3) months of the simulation experience.
  Interventions: Other: simulation based learning

INTERVENTIONS:
Other: simulation based learning — An educational methodology that aims to improve participants' attitudes towards the elderly and their perception of individualized care.

SUMMARY:
The elderly population is increasing in the world. Therefore, it is necessary to competent nurses who can diagnose the care needs of the elderly. Trainings should be planned in order to improve nurses' perception of individualized care in the care and attitudes positively of elderly patient. In post-graduate education, the use of traditional teaching methods and innovative simulation-based education will facilitate the increase of knowledge and skills. The aim of this study is to examine the effect of simulation-based education on the improve of nurses' perception of individualized care and positive attitudes towards the elderly. The study is quasi-experimental with a pre-test post-test design. Before the data collection phase, a simulation-based training program consisting of three stages was created. The data of the study were collected in a university hospital between October 2021 and April 2022, with the socio-demographic characteristics form, the perception of individualized care and the attitude scale towards the elderly. The data will be analyzed in the package program and the study will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Completed undergraduate education
* Have been working in the geriatric clinic for at least 6 months
* Volunteer to participate in the study

Exclusion Criteria:

* Not completing the stages of the study
* nurses with less than 6 months of experience in the geriatric clinic
* not volunteer to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Change from attitudes towards the elderly at four months | Pre-test (before theoretical course), post test 1 (one week after simulation-based learning), post test 2 (one month after simulation-based learning) and post test 3(three month after simulation-based learning)
  Mean scores of the participants' on scale of attitude towards the elderly
Change from perception of individualized care at four months | Pre-test (before theoretical course), post test 1 (one week after simulation-based learning), post test 2 (one month after simulation-based learning) and post test 3 (three month after simulation-based learning)
  Mean scores of the participants on the scale of perception of individualized care for the elderly
Change from knowledge test at four months | Pre-test (before theoretical course), immediately post test 1, post test 2 (one week after simulation-based learning), post test 3 (one month after simulation-based learning) and post test 4 (three month after simulation-based learning)
  Mean scores of the participants' on scale of knowledge of care towards the elderly

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study is a doctoral thesis. It will first be reported as a thesis and then shared with the researchers as an article.
Supporting Information: CSR
Time Frame: The data will be used until the thesis and article process is completed.